CLINICAL TRIAL: NCT00391404
Title: Randomized Controlled Study on the Benefits and Safety of Bisphosphonate Treatment in Childhood Cancer Survivors
Brief Title: Fosamax for Childhood Cancer Survivors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HK-CCFGrants2005.TFL
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Osteoporosis
Keywords: Childhood cancer survivors; Osteoporosis; Bone mineral density; Therapy; Bisphosphonate; Randomized controlled trial
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alendronate (Active Comparator): Oral alendronate 70 mg weekly
  Interventions: Drug: Alendronate
- Placebo (Placebo Comparator): Conventional drug treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate — Alendronate 70 mg weekly (oral)
  Other Names: Fosamax
  Arms: Alendronate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Survivors of childhood cancers face a variety of long-term problems. The investigators' recent study found that osteoporosis and osteopenia were common among these patients. The factors leading to, as well as the best treatment option for, this morbidity are unclear. Bisphosphonates are currently the standard therapy for osteoporosis in the elderly. However, the efficacy and safety of bisphosphonates for treating osteoporosis in long-term cancer survivors have not been tested. The investigators hypothesize that alendronate, an orally active bisphosphonate, is efficacious and safe in the treatment of osteoporosis in these patients.

DETAILED DESCRIPTION:
The modern treatment for childhood malignancy includes surgery and chemoradiotherapy either individually or in combination. Despite the great achievement in improving patient survival, these treatments also greatly enhance the adverse effects on the unfortunate children. Our research group has recently conducted a pioneer study on the bone mineralization and bone mineral density (BMD) study in longterm childhood cancer survivors in local patients who have completed anti-cancer treatment for at least five years. This landmark study showed that persistent treatment-related adverse effects on skeletal development are common (up to 50%) in local long-term survivors of childhood cancers. Thus, it is important during this critical period of rapid somatic growth in adolescents and young adults that these cancer survivors achieve their peak potential for bone mineralization and strengthening. In this proposed study, we investigate with a randomized and controlled study design on the efficacy of a second-generation oral bisphosphonate, alendronate, to improve BMD over a 36-week period in long-term survivors of childhood cancers in Hong Kong. In addition to alendronate, all subjects in the active and control groups will receive alfacalcidol (vitamin D) and calcium carbonate throughout the whole study period. The study results will help paediatric oncologists to decide on the optimal remedial treatments against osteoporosis in long-term cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Chinese patients who completed treatments for childhood cancers for at least 5 years
* Currently followed up in the Department of Paediatrics of Prince of Wales Hospital
* Younger than 18 years old at the time of diagnosis of underlying cancers
* Evidence of osteoporosis (i.e. BMD T- or Z-score < -2.5 at lumbar spine)
* Older than 15 years of age at the time of recruitment

Exclusion Criteria:

* Current treatment (i.e. within 6 months) with maintenance systemic or high-dose inhaled corticosteroids
* Subjects who cannot cooperate for BMD measurements
* Pregnant female patients
* Subjects with prior history of allergy to alendronate or in whom alendronate treatment is contraindicated

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
The percent change in bone mineral density (BMD) at lumbar spine at 36-weeks in subjects who receive active and control treatments | 36 weeks

SECONDARY OUTCOMES:
Changes in BMD at femoral neck | 36 weeks
Changes in biochemical markers of bone turnover | 36 weeks
Occurrence of clinical bone-related symptoms at 12-weeks and end of this study | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting Fan Leung, MBChB, MD, Principal Investigator — Department of Pediatrics, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, N.T., Hong Kong, Hong Kong